CLINICAL TRIAL: NCT02398903
Title: Pharmacological Evaluation of Hormonal Contraceptive Treatments in Obese Women Before and After Bariatric Surgery
Brief Title: Evaluation of Hormonal Contraceptive Treatments in Obese Women
Acronym: OBECO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P 130942
Record Dates: First submitted 2015-02-09; First posted 2015-03-26 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Bariatric Surgery Candidate; Oral Contraceptive
Keywords: Morbid obesity; bariatric surgery; sleeve gastrectomy; Roux-en-Y gastric bypass; hormonal contraception; combined oral contraceptive; progestin contraceptive desogestrel; pharmacokinetics
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for measurement of drug Css
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese women SG: Obese women operated by sleeve gastrectomy
  Interventions: Other: Blood samples for measurement of drug Css; Other: DXA and impedancemetry
- Normal weight women: Normal weight women
  Interventions: Other: Blood samples for measurement of drug Css; Other: DXA and impedancemetry
- Obese women GBP: Obese women operated by Rougastric bypass
  Interventions: Other: Blood samples for measurement of drug Css; Other: DXA and impedancemetry

INTERVENTIONS:
Other: Blood samples for measurement of drug Css — Blood samples for measurement of drug Css
Other: DXA and impedancemetry — Body composition by DXA and impedancemetry

SUMMARY:
The aim of our study is to assess the concentrations of different oral contraceptive agents in morbid obese women before and after two types of bariatric surgeries (RYGB and sleeve gastrectomy) in order to study the role of the surgery and the role of body weight on drug concentrations, and to compare these concentrations with those of normal-weight women.

DETAILED DESCRIPTION:
Open, multi-center pharmacological study of residual concentrations of three different oral contraceptives in 3 groups of obese women in each group of surgery, and 1 group of healthy volunteers. The concentrations will be assessed before, 6 and 12 months after bariatric surgery restrictive (sleeve gastrectomy) or malabsorptive (gastric by pass).

Contraception is an important issue in women with obesity. There are actually few data answering the questions of the efficacy of oral contraceptive in obese women, as this condition could be a risk factor for failure of hormonal contraception, due to the changes in drug metabolism and a larger volume of distribution in obesity. Bariatric surgery is the most efficient therapeutic for weight loss in severe and morbid obesity. In 2011, more than 31 000 bariatric procedures have been performed in France with sleeve gastrectomy and Roux-en-Y gastric bypass (RYGB) representing the two most frequent procedures. Women represent 80 % of surgical patients and most of them are in childbearing age (mean age of 39 years). Obese women who receive surgical treatment for obesity are advised not to conceive for the following 12 to 18 months, both to ensure optimal weight loss and a stable weight during pregnancy, and also to begin pregnancy with optimal nutritional and vitamin status. There are no data on the changes in oral contraceptives concentrations before and after bariatric surgery, as malabsorption and anatomic digestive modifications following surgery may theoretically affect bioavailability.

Primary Objective :

The difference between Css before bariatric surgery and 6 months after the surgery in obese women regardless of the oral contraceptives used. Three different oral contraceptives are employed (two combined oral contraceptive containing ethinyl E2 and levonorgestrel and a progestin contraceptive desogestrel).

Secondary Objectives :

* To assess if the difference of Css before, 6 months and 12 months after surgery is the same in the 3 groups of oral contraceptives and in the 2 groups of surgery
* To compare the Css of obese women before, 6 months and 12 months after surgery to T0 Css of normal-weight patients for each group of oral contraceptive
* To assess the impact of oral contraceptives on gonadotroph axis, hemostatic variables and estrogen-sensitive protein in obese women before and 6 and 12 months after surgery and in normal-weight women
* Analyze of correlation between body composition, nutritional status and Css in the 3 groups of oral contraceptives and in the 2 groups of bariatric surgery

Secondary End Points:

* Css of oral contraceptive agent 12 months after bariatric surgery
* Css of oral contraceptive agent in normal weight women
* Sequential Body composition by DXA and Impedancemetry before and 6 months and 12 months after surgery.
* Nutritional status in obese women before and after surgery (albumin, prealbuminemia, RBP, transferrin, haemoglobin, lipid (total cholesterol, triglycerides, LDL and HDL)
* Evaluation of gonadotroph axis by hormonal assays: FSH, LH, estradiol, AMH, progesterone, testosterone total, Inhibin B in normal-weight women and obese women before and 6 months and 12 months after surgery
* Evaluation of hemostatic variables (protein S, APC) and SHBG in normal-weight women and obese women before and 6 months and 12 months after surgery
* Number of unexpected pregnancies occurred during the study

ELIGIBILITY:
Eligibility Criteria:

Inclusion criteria :

* Obese women

  * Obese women (BMI ≥ 35 kg/m² with obesity related comorbidity or BMI ≥ 40 kg/m²) with an indication of bariatric surgery by RYGB or sleeve gastrectomy under oral contraceptive treatment of interest in our study
  * Aged 18 to 45 years if desogestrel or 18 to 35 years if COC
  * Signed informed consent
  * Affiliated to The French Social Security Health insurance
* Healthy Volunteers

  * Normal weight (BMI < 25 kg/m²)
  * Women under oral contraceptive treatment
  * Aged 18 to 45 years
  * Signed informed consent
  * Affiliated to The French Social Security Health insurance

Exclusion criteria :

* Drug treatment known to interact with cytochrome P450 (CYP3A4).
* Contraindication for an oral contraceptive agent as mentioned in the summary of product characteristics
* Positive pregnancy test

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese women with an indication of bariatric surgery by RYGB or sleeve gastrectomy under oral contraceptive treatment.
  Normal-weight women under oral contraceptive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2015-03-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Css | 6 months
  The difference between Css before bariatric surgery and 6 months after the surgery in obese women regardless of the oral contraceptives used. Three different oral contraceptives are employed (two combined oral contraceptive containing ethynil E2 and levonorgestrel and a progestin contraceptive desogestrel).

SECONDARY OUTCOMES:
Css | 12 months
  • To assess if the difference of Css before, 6 months and 12 months after surgery is the same in the 3 groups of oral contraceptives and in the 2 groups of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bachelot, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Pitié Salpetriere Hospital, Paris

IPD SHARING:
Plan to Share IPD: No